CLINICAL TRIAL: NCT03524144
Title: Upper Gastrointestinal Lesions in Crohn's Disease: a Cross-sectional Cohort Study
Brief Title: Upper Gastrointestinal Lesions in Crohn's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiang Gao, Clinical Professor, Sixth Affiliated Hospital, Sun Yat-sen University
Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2017ZSLYEC-097
Record Dates: First submitted 2018-04-30; First posted 2018-05-14 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Upper Gastrointestinal Lesions; Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Gastroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- adult patients with Crohn's disease (Other): All adult patients(18 years old or older) with Crohn's disease underwent gastroscopy; patients with diagnosed and treated Crohn's disease had gastroscopy performed during the re-examination, and patients diagnosed with Crohn's disease for the first time had gastroscopy performed during the initial consultation.
  Interventions: Other: gastroscopy

INTERVENTIONS:
Other: gastroscopy — Two endoscopists performed upper gastrointestinal endoscopy and biopsy on all patients; and histological review was performed by two pathologists. From each patient, 10 specimens were taken from 6 areas in the upper gastrointestinal tract and basic informations was collected.

SUMMARY:
A cross-sectional study was performed from 2017 to 2018. Consecutive Crohn's disease patients diagnosed in the Inflammatory bowel disease center of the Sixth Affiliated Hospital of Sun Yat-sen University were recruited. All patients underwent upper gastrointestinal endoscopy and biopsy by two defined endoscopists and two pathologists, the basic information were collected at the same time, in order to assess the prevalence of upper gastrointestinal involvement, and determine the role of upper gastrointestinal endoscopy in adult Crohn's disease patients, irrespective of upper gastrointestinal symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age is 18 years old or older
* patients with diagnosis of Crohn's disease

Exclusion Criteria:

* diagnostic data were incomplete
* patients with malignant tumor
* use of PPIs or non-steroidal anti-inflammatory drugs in the preceding 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-05-30 (Estimated); Study Completion 2018-05-30 (Estimated)

PRIMARY OUTCOMES:
the incidence of different upper gastrointestinal lesions | 1 year
  The incidence of different characteristic lesions of upper gastrointestinal in CD patients.

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Gao, Study Chair — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China